CLINICAL TRIAL: NCT03802201
Title: A Phase 2 Study of PTG-300 in Non-Transfusion Dependent (NTD) and Transfusion-Dependent (TD) β-Thalassemia Subjects With Chronic Anemia
Brief Title: Study of PTG-300 in Non-Transfusion Dependent and Transfusion-Dependent Beta-Thalassemia Subjects With Chronic Anemia
Acronym: TRANSCEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PTG-300-02
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: β-thalassemia; Ineffective Erythropoiesis; Chronic Anemia
Keywords: chronic anemia; β-thalassemia

STUDY DESIGN:
Intervention Model Description: Multiple PTG-300 dose levels/regimens are planned to be tested for each subpopulation of β thalassemia (NTD and TD) on separate arms:
  * Cohort 1: 3 mg subcutaneous (SC) weekly
  * Cohort 2: 10 mg SC weekly
  * Cohort 3: 20 mg SC weekly
  * Cohort 4a: 40 mg SC weekly
  * Cohort 4b: 40 mg SC every 2 weeks
  * Cohort 7: 80 mg SC weekly
  * Cohort 8: 40 mg SC twice a week
  Additional Cohorts (Cohorts 5,6,9,10, and 11) will include subjects between 12 years of age and less than 18 years of age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTG-300 Active (Experimental): Drug: PTG-300 Subcutaneous
  Interventions: Drug: PTG-300

INTERVENTIONS:
Drug: PTG-300 — Subcutaneous (SC)

SUMMARY:
This is a Phase 2 open-label, single-arm design study with dose escalation by subject cohort . The study is designed to monitor the PTG-300 safety profile, to obtain preliminary evidence of efficacy of PTG-300 for the treatment in β-thalassemia.

DETAILED DESCRIPTION:
This is a Phase 2 open-label, single-arm design study with dose escalation by subject cohort and with the potential for individual titration (dose increase or decrease) within each cohort. The study is designed to monitor the PTG-300 safety profile, to obtain preliminary evidence of efficacy of PTG-300 for the treatment of chronic anemia in β-thalassemia and to evaluate the appropriate dosing regimen for PTG-300 in the target population

ELIGIBILITY:
Main Inclusion Criteria:

1. Male and female subjects aged 18 to 65 years, inclusive (Cohorts 1-4b).
2. Male and female subjects aged 12-<18 years, with a minimum weight of 30 kg (Cohorts 5 and 6).
3. Documented diagnosis of β-thalassemia with no other Hgb abnormality.

Inclusion criteria applicable only for NTD β-thalassemia subjects:

1. Mean Hgb < 10.0 g/dL of two measurements (one performed 7-28 days prior to dosing and the other performed within 7 days prior to dosing).
2. Requirement of < 6 units RBC transfusion in a 24 week period with the last transfusion at least 8 weeks before screening.

Inclusion criteria applicable only for TD β-thalassemia subjects:

1. Transfusion requirement of at least 6 units of RBC in the 24 weeks prior to screening with no transfusion free period > 45 days.
2. Last RBC transfusion 5-10 days prior to dosing.

Main Exclusion Criteria:

1. Subjects with Sickle Cell disease, Hgb H, Hb Bart's hydrops foetalis or hemoglobin S
2. Infection requiring hospitalization or IV antimicrobial therapy, or opportunistic infection within 6 months of dosing, any infection requiring antimicrobial therapy within 2 weeks of dosing; history of infection with human immunodeficiency virus (HIV).
3. Subject has a concurrent clinically significant, unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic or other medical disorder that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the subject by their participation in the study.
4. Known primary or secondary immunodeficiency.
5. History within 6 months of screening of any of the following:

   myocardial infarction, unstable angina, transient ischemic attack, decompensated heart failure requiring hospitalization, congestive heart failure (New York Heart Association Class 3 or 4), uncontrolled arrhythmias, cardiac revascularization, stroke, uncontrolled hypertension (resting systolic blood pressure [BP] > 160mmHg or resting diastolic BP > 100mmHg on more than one occasion) or uncontrolled diabetes (Hgb A1c > 9% or > one episode of severe hypoglycemia).
6. Pregnant or lactating females.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
NTD: Proportion of responders at each dose | 4 week period
  NTD subjects who achieve an increase in Hgb without transfusion
TD: Proportion of clinical responders at each dose | 8 week period
  TD subjects who achieve a reduction in red blood cell (RBC) units required over an 8 week period

CONTACTS AND LOCATIONS:
Locations (32):
- United States (3):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
- Greece (4):
  - University General Hospital of Patras, Pátrai, Achaia
  - Laiko General Hospital of Athens, Athens, Attica
  - Athens General Hospital 'G Gennimatas', Athens, Attica
  - Hippokration Hospital, Thessaloniki
- Italy (3):
  - Presidio Ospedaliero Antonio Perrino, Brindisi
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Napoli
- Chronic Care Center, Beirut, Lebanon
- Malaysia (5):
  - Hospital Ampang, Ampang
  - Hospital Pulau Pinang, George Town
  - Hospital Sultanah Aminah, Johor Bahru
  - Queen Elizabeth Hospital, Kota Kinabalu
  - Hospital Umum Sarawak, Kuching
- Thailand (5):
  - Chulalongkorn University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Naresuan University, Phitsanulok
- Tunisia (4):
  - University Hospital Farhat Hached, Sousse
  - Bone Marrow Transplant Center, Tunis
  - Aziza Othmana Hospital, Tunis
  - Principal Military Hospital, Tunis
- Turkey (Türkiye) (6):
  - Acibadem Adana Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Mersin University Medical Facult, Mersin
- Barts Health NHS Trust, London, United Kingdom